CLINICAL TRIAL: NCT03704909
Title: Managing Post Spinal Hypotension During Elective Cesarean Section: Epinephrine Versus Ephedrine, a Randomized Double-blinded Controlled Trial
Brief Title: Manging Post Spinal Hypotension During Elective Cesarean Section
Acronym: EpiEph
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ben marzouk Sofiene (Other)
Responsible Party: Sponsor-Investigator, Ben marzouk Sofiene, clinical associate professor, University Tunis El Manar
Organization: University Tunis El Manar (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Adrenaline
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Hypotension
Keywords: Epinephrine, Ephedrine, cesarean section, spinal anesthesia
MeSH Terms: conditions — Hypotension | interventions — Epinephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Adrenaline: Group A (Active Comparator): All parturients received a prophylactic i.v bolus of Epinephrine 0.15µg/Kg at time of SA. In this group, rescue boluses of Epinephrine 0.15µg/Kg, will be given if maternal BP decreased more than 20% from the baseline value.
  Interventions: Drug: Adrenaline
- Group Ephedrine: Group E (Active Comparator): All parturients received a prophylactic i.v bolus of Ephedrine 0.1mg/Kg at time of SA. In this group, rescue boluses of Ephedrine 0.1mg/Kg, will be given if maternal BP decreased more than 20% from the baseline value.E
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Adrenaline — i.v bolus of adrenaline 0.15µg/Kg rescue boluses of adrenaline 0.15µg/Kg
  Other Names: epinehrine
  Arms: Group Adrenaline: Group A
Drug: Ephedrine — i.v bolus of Ephedrine 0.1mg/Kg rescue boluses of Ephedrine 0.1mg/Kg
  Arms: Group Ephedrine: Group E

SUMMARY:
Spinal anesthesia is the gold standard technique for elective cesarean section. It helps to avoid risks regarding airway management and provides effective neuraxial postoperative analgesia, enabling quicker maternal recovery. Cesarean section normally require an anesthetic block at T4 level. So that maternal hypotension is reported to occur in up to 80%. This can result in significant morbidity for both the mother and fetus.The purpose of this study is to determine if epinephrine is as effective and safe compared to ephedrine for maintaining arterial blood pressure during elective cesarean section under spinal anesthesia. All participants will receive spinal anesthesia with a local anesthetic and sufentanil. This study plans to enroll 140 healthy pregnant women. Patients will be randomly assigned according to a computer generated system to be in one of two groups.

DETAILED DESCRIPTION:
Its a prospective double-blinded controlled trial. All participants gave a written informed consent. One hundred and twenty healthy women, ASA II, with singleton pregnancies at term scheduled for elective cesarean section under spinal anesthesia are targeted for the study. They are randomized to receive either epinephrine or ephedrine. Upon arrival in the operating room, parturient was placed in the supine position with 15° left lateral tilt with routine monitoring (HR, non-invasive BP, pulse oximetry, electrocardiography). Baseline BP and HR were computed as the mean of three consecutive BP and HR readings respectively at 1-minute intervals. Study participants will receive a standard spinal anesthetic consisting of 0.5% hyperbaric bupivacaine (2 mL) plus sufentanil (5 µg) at L3-4 vertebral interspace.

Group A (for adrenaline group): received a prophylactic intravenous (i.v) bolus of Epinephrine 0.15µg/Kg at time of SA. In this group, rescue boluses of Epinephrine 0.15µg/Kg, were given if maternal BP decreased more than 20% from the baseline value.

Group E (for ephedrine group): received a prophylactic i.v bolus of Ephedrine 0.1mg/Kg at time of SA. In this group, rescue boluses of Ephedrine 0.1mg/Kg, were given if maternal BP decreased more than 20% from the baseline value. Once the spinal injection was performed a rapid intravenous (i.v.) coload with 15mL/Kg of isotonic saline solution was started through a 16 G i.v. cannula (by turning the i.v. infusion to maximum and using a pressure bag inflated to 150 mmHg). A prophylactic bolus of vasopressor was administered at the end of spinal injection. After performing anesthesia, the parturient was immediately replaced in the supine position with a 15° left lateral table tilt until delivery of the infant. Prior to surgical incision, the spinal sensory level will be tested to the bilateral T6-T4 dermatomal level. Sensory block level was checked by cold-hot test and the Modified Bromage Scale was used for the assessment of motor block. The surgery was allowed when the sensory block level reached D4. Both the patient and the researcher's assistant (who will collect data) will be blinded as to the administered Epinephrine or Ephedrine bolus. Supplemental oxygen will be given only when the pulse oximeter reading decreased below 95%. After delivery, 5 IU of oxytocin diluted in 20 ml of isotonic saline solution were slowly injected over 1 minute. Then an i.v infusion was given (10 IU/500ml of isotonic saline solution at a flow rate of 28 drops/min).

Heart rate (beats/min), systolic, mean and diastolic blood pressure (mmHg) will be recorded every 1 min after spinal injection until the end of surgery. The incidence of hypotension (defined as a reduction in SBP of >20% from baseline determined just before the administration of spinal anesthesia) will be recorded. Reactive hypertension (defined as a rise of SBP >20% of baseline) will also be recorded. Bradycardia (defined as HR <50 beats/min) will be recorded. Tachycardia (defined as a HR >140 beats/min) will also be recorded. Umbilical blood samples will be obtained by clamping it on both sides and a gas analysis will be performed to determine fetal pH, HCO3-, base excess and lactates. Furthermore, Apgar scores at 1 and 5 minutes after delivery will be recorded by the attending pediatrician, who will be unaware of the vasopressor used. The study will end when cesarean section is completed and the patient is transferred to the post-operative care unit.

ELIGIBILITY:
Inclusion Criteria:

* ASA II
* BMI>18 and <35 Kg/m2
* full term parturients with singleton pregnancy
* scheduled of elective cesarean section under spinal anesthesia

Non-inclusion criteria:

* Patient refusal.
* ASA > II
* Preexisting or pregnancy-induced hypertension
* The use of cardiac medication or medication for BP control.
* Cardiovascular or cerebrovascular disease.
* Multiple pregnancy.
* Suspicion of abnormal placentation.
* Known fetal abnormalities or fetal distress.
* CS under general anesthesia.
* Active labor.
* Emergency.
* Allergy to any of the medications used in the study.

Exclusion Criteria:

* Hemodynamic instability that is not in relationship with SA (occurrence of a surgical per-operative complication e.g. bleeding by placental insertion abnormality or a uterine atony).
* An abnormal extension of the anesthetic block defined as a sensory block level > D4.
* SA failure.
* The need to convert to general anesthesia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
delta SBP (D) | at the end of intrathecal injection until delivery
  difference between baseline and the lowest systolic blood pressure.
delta MBP (D) | at the end of intrathecal injection until delivery
  difference between baseline and the lowest mean blood pressure.

SECONDARY OUTCOMES:
delta SBP (S) | at the end of intrathecal injection until the end of surgery
  difference between baseline and the lowest systolic blood pressure.
delta MBP (S) | at the end of intrathecal injection until the end of surgery
  difference between baseline and the lowest mean blood pressure.
time to onset of first post spinal hypotension episode | At time of surgery (right after spinal anesthesia until end of surgery)
  first episode of hypotension after spinal anesthesia induction
Incidence of post spinal hypotension | At time of surgery (right after spinal anesthesia until end of surgery)
  a decrease of SBP >20% of baseline
Vasopressor consumption | from the end of intrathecal injection until delivery.
  cumulative dose of vasopressor consumption
Vasopressor consumption | from the end of intrathecal injection until the end of surgery.
  cumulative dose of vasopressor consumption
number of rescue boluses | At time of surgery (right after spinal anesthesia until end of surgery)
  number of rescue boluses before and after delivery
incidence of hypertension | At time of surgery (right after spinal anesthesia until end of surgery)
  a rise of SBP >20% of baseline
tachycardia | At time of surgery (right after spinal anesthesia until end of surgery)
  heart rate>140 beats/min
incidence of arrythmia | At time of surgery (right after spinal anesthesia until end of surgery)
  incidence of arrhythmic events
incidence of bradycardia | At time of surgery (right after spinal anesthesia until end of surgery)
  heart rate (HR) < 50 beats/min
use of atropine | At time of surgery (right after spinal anesthesia until end of surgery)
  cumulative dose, if needed
incidence of nausea and vomiting | At time of surgery (right after spinal anesthesia until end of surgery)
  Measure will be done according to a simple scale: 0= no nausea and vomiting; 1= nausea or vomiting
foetal gas analysis: pH, Lactates, HCO3-, BE | At time of birth
  fetal cord blood analysis will be done immediately after delivery
APGAR score | at 1 and 5 minutes after birth
  range from 0 to 10,incorporates five elements: respiratory effort, heart rate, reflex irritability, muscle tone, and color A score of 0 to 3 indicates a severely depressed neonate, whereas a score of 7 to 10 is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: HAYEN MAGHREBIG, PROFESSOR, Study Chair — UNIVERSITY OF TUNIS EL MANAR
Locations (1):
- Tunis maternity and neonatology center,, Tunis, Tunisia